CLINICAL TRIAL: NCT04832373
Title: Assessment of the Acceptability of a Humanoid Robot at Home for Children With Cochlear Implants - H2R2
Acronym: H2R2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0250; 2020-A01989-30. (Other: ID-RCB)
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-02

CONDITIONS: Cochlear Implantation
Keywords: cochlear implantation; humanoid robot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Humanoid Robot (Other)
  Interventions: Device: Interaction with humanoid robot

INTERVENTIONS:
Device: Interaction with humanoid robot — A humanoid robot will be installed for 30 days in children. It has a touchscreen tablet, allowing manual interaction complementing the voice interaction. The robot speaks, hears, and has facial and voice identification.

SUMMARY:
The quality of the rehabilitation of deafness in children with cochlear implantation is a major prognostic factor for the outcome on speech comprehension and oral expression. This rehabilitation is carried out cooperatively by the hospital cochlear implantation team, and by a speech therapist located near the child's home. The multi-weekly sessions represent a constraint for the child and his parents. Complementary training work at home would make it possible to balance the equity in the distribution of care in the territory, and should promote the progress of the child, who is more inclined to use a tool available at home.

DETAILED DESCRIPTION:
The humanoid robot should allow an ecological approach to this additional rehabilitation. Before developing this approach, it is necessary to study the acceptability of the humanoid robot at home, both by the parents and by the cochlear implanted child. The main objective of this study is to assess the acceptability by the child and his family, of a humanoid robot installed at home for one month.

The secondary objectives are to describe the acceptability of the child and his family that is the relationship to technology, the intention of use, expectations, perceived utility, perception of the robot and facilitating conditions before then after 1 month of using the robot at home,

- describe the child's acceptability with respect to his experience, his fun and the emotions felt when he uses the robot at home

ELIGIBILITY:
Inclusion Criteria:

* Child aged 8 to 12, user of his cochlear implant with a favorable family environment,
* Child implanted with at least one cochlear implant undergoing speech therapy rehabilitation, and monitored by the pediatric cochlear implant unit (UPIC) of the Toulouse University Hospital
* Child and his family whose mother tongue is French
* Affiliation to a social security scheme

Exclusion Criteria:

* Cognitive or psychological inability or refusal of the participant to give written consent
* Other sensory or motor deficit that may interfere with the use of the robot
* Unstable psychiatric pathology
* Child with both parents benefiting from a legal protection measure

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Acceptability of a humanoid robot | month 1
  assess by the number of weekly hours during which the child uses the robot.

SECONDARY OUTCOMES:
Relationship to technology | month 1
  Assessment by a set of questionnaires and standardized scales validated by the scientific community
Intention of use | month 1
  Assessment by a set of questionnaires and standardized scales validated by the scientific community
Relationship with the robot | month 1
  Assessment by a set of questionnaires and standardized scales validated by the scientific community
User experience | Month 1
  Assessment by a set of questionnaires and standardized scales validated by the scientific community
participants' expectations | Month 1
  Measurement by sentence completion which consists of giving the beginning of a sentence and letting the user complete the rest of the sentence
3Emethod | Month 1
  Evaluation of emotions in the form of a drawing with a speech bubble and a thought bubble.
classification of activities | Month 1
  classification according to various criteria (good functioning, fun, ease of use)
Feedback | Month 1
  with a Semi-structured interview on the use of the robot

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DEGUINE, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse - Service d'ORL, ORL pédiatrique et Otoneurologie, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stiti S, Caroux L, Gaillard P, Paubel PV, Deguine O. Innovative protocol of an exploratory study evaluating the acceptability of a humanoid robot at home of deaf children with cochlear implants. PLoS One. 2023 Jun 16;18(6):e0285927. doi: 10.1371/journal.pone.0285927. eCollection 2023. PMID 37327230
- [Background] Diehl JJ, Schmitt LM, Villano M, Crowell CR. The Clinical Use of Robots for Individuals with Autism Spectrum Disorders: A Critical Review. Res Autism Spectr Disord. 2012 Jan;6(1):249-262. doi: 10.1016/j.rasd.2011.05.006. PMID 22125579